CLINICAL TRIAL: NCT05389007
Title: German TTP- Registry- Prospective Cohort of Patients With Acquired Thrombotic Thrombocytopenic Purpura (aTTP): Pathophysiology, Diagnosis, Treatment and Follow-Up
Brief Title: .German TTP-Registry (Thrombotic Thrombocytopenic Purpura)
Acronym: RGTTP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Charis v. Auer, Head of Hemostaseology, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: RGTTP
Record Dates: First submitted 2022-05-09; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Open, multi-center, observational, prospective cohort study, only disease-indicated treatment, in patients with clinically diagnosed acquired and congenital TTP regardless of gender, ethnicity, and comorbidities, over the age of 18 for 1.) prospective investigation of patients with TTP in an acute bout and during long-term follow and 2.) assessment of prevalence, course of disease, success of therapy, possible triggers for relapses and possibilities for better diagnosis and prognosis.

DETAILED DESCRIPTION:
1.) Identification of predictive markers for morbidity and mortality in acute TTP and in TTP relapses using a prospective long-term registry and 2.) Investigation of the pathophysiological processes in acute bouts and in remission by recording the clinical symptoms and diagnostics for a better understanding of the course of the disease, optimization of diagnostic procedures and their correlation with the clinical course, recording of therapy response of all therapeutic options in acute bouts, observation of current treatment options to evaluate outcome and prognostic markers and recording of clinical and laboratory chemical data during follow-up to assess long-term morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed acquired and congenital TTP regardless of gender, ethnicity, and comorbidities, over the age of 18.
* Patients incapable to give consent, who are accompanied by a legal representative during admission to the study, after the written informed consent of the legal representative.
* Written informed consent of the patient.

Exclusion Criteria:

* Patients who are not able to understand the German or English language.
* Patients who are permanently unable to communicate and who are not accompanied by a legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include all patients with TTP in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 156
Dates: Start 2016-07-08; Primary Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Predictive markers for morbidity and mortality | 3 years
  Identification of predictive markers for morbidity and mortality in acute TTP and in TTP relapses using a prospective long-term registry

CONTACTS AND LOCATIONS:
Overall Officials: Charis v. Auer-Wegener, Principal Investigator — Universitätsmedizin Mainz
Locations (1):
- University Hospital Mainz, Hematology, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No